CLINICAL TRIAL: NCT01365715
Title: Preoperative Embolization in Surgical Treatment of Spinal Metastases. A Randomized Controlled Trial.
Brief Title: Preoperative Embolization in Surgical Treatment of Spinal Metastases.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Caroline Clausen, MD, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H-2-2011-024; H-2-2011-024 (Other: The Danish Committee on Biomedical Research Ethics); 2008-41-2128 (Other: Danish Dataprotection Agency)
Record Dates: First submitted 2011-05-27; First posted 2011-06-03 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-02

CONDITIONS: Spinal Metastases
Keywords: Preoperative embolization; Transcatheter arterial embolization; Therapeutic angiography; Embolization; Surgical blood loss; Spinal metastases; Spinal neoplasms; Vertebral metastases; metastatic spine surgery; Spinal surgery
MeSH Terms: conditions — Blood Loss, Surgical; Spinal Neoplasms | interventions — Embolization, Therapeutic; Cerebral Angiography

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Preoperative embolization (Experimental): 32 patients with spinal metastasis/metastases will undergo arteriography and receive transcatheter arterial embolization of spinal metastasis/metastases 0-48 hours prior to surgery.
  Interventions: Procedure: Arteriography and preoperative embolization
- Control group (Active Comparator): 32 patients with spinal metastasis/metastases will undergo arteriography of spinal metastasis/metastases without receiving transcatheter arterial embolization prior to surgery.
  Interventions: Procedure: Arteriography

INTERVENTIONS:
Procedure: Arteriography and preoperative embolization — Arteriography and transcatheter arterial embolization of spinal metastasis/metastases 0-48 hours prior to surgery.
  Other Names: Transcatheter arterial embolization; Selective arterial embolization; Therapeutic angiography; Embolization
  Arms: Preoperative embolization
Procedure: Arteriography — Arteriography of spinal metastasis/metastases without transcatheter arterial embolization prior to surgery.
  Other Names: Angiography
  Arms: Control group

SUMMARY:
The main purpose of this study is to assess the efficacy of preoperative embolization in decreasing operative blood loss, decreasing the need for intraoperative transfusion and facilitate surgical resection in metastatic spine surgery. Furthermore the study aims at describing the vascularity in a series of spinal metastasis, and to correlate this with perioperative blood loss.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for decompression and posterior thoracic and/or lumbar instrumented spinal fusion because of spinal metastasis/metastases.
* Informed signed consent.

Exclusion Criteria:

* Contrast fluid allergy.
* Clotting disorders.
* Renal failure.
* Not suitable for arterial access.
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2011-05; Primary Completion 2014-02 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
Perioperative blood loss | Measured intraoperatively and 24 hours postoperatively.

SECONDARY OUTCOMES:
Perioperative blood transfusion volume | Intraoperatively and until 48 hours postoperatively.
Surgical procedure time. | At skin closure.
  Defined as the amount of time (measured in minutes) from skin incision to skin closure.
Vascularization grade of metastasis | At the angiographic procedure prior to embolization performed 0-48 hours before surgery.
Success of embolization | Directly after the embolization performed 0-48 hours before surgery.
Adverse events related to angiography or embolization | Within 2 postoperative days
Adverse events related to surgery | Within 2 postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lönn, MD, Ph.d., Study Chair — Department of Radiology, Rigshospitalet. Copenhagen, Denmark.
Locations (1):
- Department of Radiology, Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- See also: Related Info — http://www.rigshospitalet.dk